CLINICAL TRIAL: NCT07017946
Title: A Pilot Trial to Investigate the Safety and Efficacy of Intestinal Microbiome Transplant (MTT) in People With Amyotrophic Lateral Sclerosis
Brief Title: Intestinal Microbiome Transplant in ALS
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00118099
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-06

CONDITIONS: Amyotrophic Lateral Sclerosis ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: All participants receive the investigational product.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MTP-101C administration (Experimental): MTP-101C is a freeze-dried encapsulated universal donor microbiome-based formulation. Participants will ingest 2 capsules daily for 3 days then 1 capsule daily. This is preceded by antibiotic conditioning with a combination of vancomycin and neomycin, followed by a bowel purgative with magnesium citrate depending upon underlying comorbidities.
  Interventions: Drug: MTP-101C

INTERVENTIONS:
Drug: MTP-101C — MTP-101C is a freeze-dried encapsulated formulation of fecal microbiota purified from the stool of healthy donors.

SUMMARY:
This is a 24-week study of intestinal microbiome transplant in people with ALS. All participants will be evaluated clinically in person for 4 visits. Blood and mailed/ fresh stool samples will also be collected. Blood samples will be used to determine changes in neurofilament light chain over time. Stool samples will be processed for microbiome analysis. Participants will have phone visits to further evaluate safety and tolerability. They will then undergo antibiotic conditioning and a standard bowel preparation before being assigned to the investigational product, MTP-101C .

DETAILED DESCRIPTION:
This is a 24-week Phase I/II study of MTT in people with Amyotrophic Lateral Sclerosis. All participants will be evaluated clinically in person at weeks 0, 4, 12, and 24 visits. Blood and mailed/ fresh stool samples will be collected at weeks 0, 4, 8, 12, and 24. Blood samples will be used to determine changes in neurofilament light chain over time. Stool samples from weeks 0, 4,8, 12, and 24 will be processed by molecular methods (metagenomics and metatranscriptomics) for microbiome analysis. Participants will also have phone visits at weeks 1, 8, 16, and 20, which will be used to further evaluate safety and tolerability and the ALSFRS-R score.

Participants will first undergo antibiotic conditioning with oral vancomycin 250 mg twice daily for 10 days. Neomycin 500 mg twice daily will be added to the last 3 days of vancomycin. This will be followed by ingestion of a standard bowel preparation with magnesium citrate. Participants will then ingest 2 capsules of MTP-101C daily for 3 days, then 1 capsule of MTP-101C daily for 8 weeks.

All participants will be assigned to the investigational product.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ALS according to Gold Coast Criteria
* Age: 18+ years at enrollment
* Fast-progressing (ALSFRS-R change of at least 1.5 points per month between last 2 measurements at screening)
* Modestly but not severely affected (ALSFRS-R score at or above 24 at screening)
* Able to swallow capsules and expected to be able to for the duration of the trial (ALSFRS-R "swallowing" score of 3 or 4 at screening)
* Expected to survive for the duration of the trial
* Taking any combination of riluzole, edaravone, and/or tofersen at a stable dose for 30 days prior to screening, or not taking any of these and not expected to during the study.
* Capable of giving written consent.
* If sexually active, must agree to use contraceptive or abstinence for duration of treatment.
* Females of child-bearing age must have negative pregnancy test at screening.

Exclusion Criteria:

* Concurrent illness or laboratory abnormalities that could confound the measurement of ALS progression or the microbiome or interfere with the ability to complete the study.
* Taking probiotics, nutraceuticals, or herbal remedies within 2 weeks of screening
* Taking antibiotics within 3 months of screening.
* Taking any investigational study drug within 30 days of screening or five half-lives of the prior agent.
* Previous exposure to MTT.
* Pregnancy.
* Known specific food allergy with anaphylaxis
* Other co-morbid conditions that, in the opinion of the study investigator, place the participant at increased risk of complications, interfere with study participation or compliance, or confound study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-27 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
ALS Functional Rating Scale, Revised (ALSFRS-R) | Weeks 0, 4, 8, 12, 16, 20 and 24
  The ALSFRS-R is a quickly administered (five minute) ordinal rating scale (ratings 0-4) used to determine patients' assessments of their capability and independence in 12 functional activities. The total score ranges from 0 to 48, where higher scores indicate better function.
ALS Quality of Life (ALSAQ-5) | Weeks 0, 4, 12, and 24
  The overall ALSAQ-5 score ranges from 0 (best imaginable health state) to 100 (worst imaginable health state).
Neurofilament Light Chain levels | Weeks 0, 4, 12 and 24
  Neurofilament light chain levels are elevated in the spinal fluid and the blood of patients with ALS and other neurodegenerative diseases, and higher levels predict more severe disease progression.
The Gastrointestinal Symptom Rating Scale (GSRS) | Weeks 0, 4, 12, and 24
  The Gastrointestinal Symptom Rating Scale (GSRS) is a 15-item questionnaire that can be used weekly to assess the severity of gastrointestinal symptoms experienced over the past week. The GSRS is designed to evaluate symptoms associated with common gastrointestinal disorders, such as reflux, abdominal pain, indigestion, diarrhea, and constipation. The questionnaire uses a seven-point Likert-type scale, with 1 representing no symptoms and 7 representing very troublesome symptoms. Higher scores on the subscales indicate more discomfort.

SECONDARY OUTCOMES:
Microbiome composition | Screening/Baseline, Week 4, Week 12, and Week 24
  Participants will also be sent collection kits to collect intestinal samples and return by mail. Data analyses will be performed to study the microbiome composition before and during the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bedlack, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No